CLINICAL TRIAL: NCT04103073
Title: Assessment Respiratory and Submental Muscles Activity During Inspiratory and Expiratory Maneuver in Patients With Obstructive Sleep Apnea Syndrome
Brief Title: Respiratory and Submental Muscles Activity During Inspiration and Expiration in Obstructive Sleep Apnea Syndrome
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Haluk TEKERLEK, Research assistant, Hacettepe University
Other Study IDs: osasemg
Record Dates: First submitted 2019-09-21; First posted 2019-09-25 (Actual); Last update posted 2022-01-20 (Actual); Status verified 2022-01

CONDITIONS: Obstructive Sleep Apnea
Keywords: obstructive sleep apnea; emg; inspiratory muscles; expiratory muscles
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study group: The patient with OSAS 35-70 years of age, clinically stabile, symptoms such as snoring, breathing cessations, and daytime sleepiness, and polysomnographic evidence consistent with mild (5<apnea hypopnea index (AHI)< 15) to moderate (16 < AHI < 30) OSAS.

SUMMARY:
In this study respiratory and submental muscle activities during during inspiratory and expiratory breathing maneuver at specific workloads will be assessed according to inspiratory and expiratory muscle strength of each obstructive sleep apnea syndrome (OSAS) patient's.

DETAILED DESCRIPTION:
Recurrent upper airway obstruction, apnea-hypopnea events, arousals and asphyxia during sleep increase the respiratory workload in patients with OSAS. This results in chronic overload of the inspiratory muscles -especially the diaphragm- and respiratory muscle fatigue in OSAS. When the literature was checked, there was no study assessing and comparing the activities of M. genioglossus, submental muscles (upper airways dilator muscles) and diaphragm during inspiration and expiration in a workload. Differences in the activity of these muscles according to the type of respiratory maneuver will provide more appropriate respiratory muscle training in patients.

ELIGIBILITY:
Inclusion Criteria:

* Between 35-70 years old
* Diagnosed with mild-moderate OSAS
* Clinically stabile

Exclusion Criteria:

* Anatomical obstructive upper airway
* Occupations that lead to sleep deprivation or alterations in the sleep-wake cycle.
* Comorbidities such as chronic obstructive pulmonary disease, asthma, interstitial lung diseases, neuromuscular diseases and psychiatric diseases

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with OSAS who will be referred to the Cardiopulmonary Rehabilitation Unit of the Faculty of Physical Therapy and Rehabilitation of Hacettepe University by Dışkapı Yıldırım Beyazıt Educational and Research Hospital Department of Chest Diseases will be included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2019-09-16 (Actual); Primary Completion 2021-09-14 (Actual); Study Completion 2021-12-14 (Actual)

PRIMARY OUTCOMES:
Pulmonary function test | about thirty minutes
  Pulmonary function will be assessed with a portable spirometer thorough the standard procedures. Pulmonary function test results will be recorded during the inspiratory and expiratory maneuver.
Respiratory muscle strength | about thirty minutes
  Respiratory muscle strength will be measured with a respiratory pressure meter. Maximal inspiratory pressure and expiratory pressure were recorded.
Surface electromyographic (sEMG) measurement of submental muscles and diaphragm | about thirty minutes
  Surface electromyographic (sEMG) activity of the submental muscle group (including the anterior belly of the digastric, mylohyoid, geniohyoid, and platysmas) and diaphragm will be measured during inspiratory and expiratory maneuver.

CONTACTS AND LOCATIONS:
Overall Officials: Haluk Tekerlek, MSc, Principal Investigator — Hacettepe University
Locations (1):
- Hacettepe University, Faculty of Pyhsical Therapy and Rehabilitation, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wheeler KM, Chiara T, Sapienza CM. Surface electromyographic activity of the submental muscles during swallow and expiratory pressure threshold training tasks. Dysphagia. 2007 Apr;22(2):108-16. doi: 10.1007/s00455-006-9061-4. Epub 2007 Feb 10. PMID 17294298